CLINICAL TRIAL: NCT06313281
Title: Effectiveness of Preoperative Antiseptic Preparation in Transnasal Skull Base Surgery: A Randomized Three-Arm Controlled Trial
Brief Title: Effectiveness of Preoperative Antiseptic Preparation in Transnasal Skull Base Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Sarah Basindwah, Neurosurgery resident, King Saud University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: E-18-3331
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Meningitis and Sinusitis in Transnasal Surgery
Keywords: Antisepsis; Skull Base; Sinusitis; Meningitis
MeSH Terms: conditions — Meningitis; Sinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): External 0.9% NaCl nasal preparation
  Interventions: Procedure: Preoperative Antiseptic preparation prior to transnasal skull base surgery
- Group 2 (Active Comparator): External nasal preparation with antisepsis by CHG 0.05%
  Interventions: Procedure: Preoperative Antiseptic preparation prior to transnasal skull base surgery
- Group 3 (Active Comparator): Intranasal irrigation with 80 mg of gentamicin added to 1000 ml of 0.9% NaCl plus external nasal preparation with antisepsis by CHG 0.05%
  Interventions: Procedure: Preoperative Antiseptic preparation prior to transnasal skull base surgery

INTERVENTIONS:
Procedure: Preoperative Antiseptic preparation prior to transnasal skull base surgery — The patient received one of three antiseptic preparation before transnasal skull base surgery

SUMMARY:
Objective: Transnasal skull-base surgery is a complex and invasive procedure that involves the use of preoperative antiseptic preparations. However, evidence supporting their use in preventing postoperative infectious complications is limited. The aim of this study is to assess the efficacy of preoperative antiseptic techniques in reducing postoperative infectious complications within 30 days of surgery.

Methods: A multicenter, prospective, randomized, single-blind, three-arm trial was conducted from February 2019 to October 2021. Participants were randomized to either of three antiseptic preparation techniques: external 0.9%NaCl nasal preparation, external 0.05% chlorhexidine gluconate, or intranasal irrigation with 80 mg of gentamicin added to 1000 ml of 0.9%NaCl plus external nasal preparation with chlorhexidine gluconate 0.05%. A total of 130 adults with skull-base pathologies were randomized, 12 were excluded before randomization for failure to meet inclusion criteria (n=9) or refusal to participate (n=3). The investigators excluded patients with evidence of infection adjacent to the surgical site, allergies to preparation methods, those who underwent craniotomy during the same admission, and pediatric patients.

DETAILED DESCRIPTION:
Study Design This is a multicenter, prospective, randomized, single-blind, three-arm trial conducted at three skull base centers in Riyadh, Saudi Arabia. The null hypothesis was that infectious outcomes would not differ between the three intervention groups.

Ethics Consideration The patients provided written informed consent to participate, and the institutional review boards approved the study of the participating institutions. This study was approved by the Ethics Review Boards (E-18-3331). This study was conducted using the CONSORT guidelines.7

Population Patients were screened at neurosurgery service in three skull base centers from February 2019 to September 2021; follow-up was completed in October 2021. Eligible patients were adults with skull base pathologies scheduled for ETSBS. The exclusion criteria included pediatric patients aged <14 years, known allergy to CHG or gentamicin, evidence of infection at or adjacent to the operative site prior to surgery, open craniotomy during hospitalization, and immunosuppression. Fourteen years of age was used as the age limit as this is the age of the pediatric population in the Saudi health system.

Interventional Groups Three antiseptic preparation techniques were utilized in this study in a stepwise fashion, from minimal to maximal antisepsis: Group 1, external 0.9% NaCl nasal preparation; Group 2, external nasal preparation with antisepsis by CHG 0.05%; and Group 3, intranasal irrigation with 80 mg of gentamicin added to 1000 ml of 0.9% NaCl plus external nasal preparation with antisepsis by CHG 0.05%

Randomization Procedure Patients were randomized into blocks of three intervention groups and distributed to the participating centers. The primary surgeon was blinded to the intervention method until the day of surgery. The patients were randomized using a computer-generated list of random numbers (http://www.randomizer.org). Block randomization in three-patient blocks based on the institution was performed to ensure that approximately equal numbers of patients in each group from each site were randomized.

Perioperative Intravenous Antibiotic Protocol One dose of preoperative intravenous antibiotics (cefazolin 1-2 g or ceftriaxone 1-2 g for most patients or vancomycin 15 mg/kg for patients allergic to cephalosporin) was administered within 60 min before the start of surgery. For postoperative antibiotics, three doses of the same antibiotic were administered if no lumbar drain was inserted. When a lumbar drain or an external ventricular drain was inserted, antibiotics were administered until the drain was removed.

Study Outcome The study's primary endpoint was the difference in the incidence of postoperative infections within 30 days of surgery between the three interventional groups. The investigators defined infections as any CNS or sinonasal infections confirmed by clinical or laboratory testing within 30 days post-surgery.

CNS infections CNS infections were defined as clinical signs of CNS infection with biochemical and/or microbiological evidence of infection. In cases of infection, biochemical markers, organism cultures, and outcomes were recorded.

Sinonasal infections Sinusitis: Acute bacterial sinusitis was defined, according to EPOS 2020 guideline definition 8, as the presence of three or more of the following: (1) nasal congestion based on patient reports or physical examination; (2) purulent nasal discharge based on patient reports or physical examination; (3) facial pressure, pain, or headache; and (4) antibiotics prescribed by a provider to treat sinusitis.

Patient Follow-Up All patients were followed up for at least 30 days postoperatively. Upon discharge, the patients were instructed to return if any signs or symptoms of infection occurred earlier than the follow-up clinical visit. They were followed up after discharge from the neurosurgery and rhinology clinics at least once within 30 days. At the end of the 30 days, the patient received a call if the clinic follow-up visit was not attended by the participant. During rhinology clinic visits, patients underwent a nasal scope examination by a rhinology attending.

Sample Size Sample size calculations were based on patient turnout and the infection rate in previous years in all three centers. With a confidence interval of 95%, and 5% as margin of error, the calculated sample size was123 patients over 24 months. This was divided into three arms of 41 patients in each intervention arm.

Statistical Analysis The data were entered and analyzed using the IBM SPSS Statistics for Windows, version 28 (IBM Corp., Armonk, N.Y., USA). Descriptive statistics such as frequencies and percentages were calculated to summarize categorical data and means and standard deviations to describe numerical variables. The chi-square test evaluated the association between the determinants and outcome variables. In contrast, the arithmetic means of continuous variables were compared using one-way analysis of variance for more than two groups. Multivariate logistic regression analysis expressed as adjusted odds ratio (AOR) and its 95% confidence interval (CI) was performed to control for the effect of confounding. Statistical significance was set at p < 0.05. Statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults with skull base pathologies scheduled for ETSBS

Exclusion Criteria:

* Pediatric patients aged <14 years
* Known allergy to CHG or gentamicin
* Evidence of infection at or adjacent to the operative site prior to surgery
* Open craniotomy during hospitalization
* Immunosuppression

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
the difference in the incidence of postoperative infections within 30 days of surgery between the three interventional groups | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrazag Ajlan, MD, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided